CLINICAL TRIAL: NCT00772785
Title: An Open-label, Multi-center Extension Study of Probuphine in Patients With Opioid Dependence
Brief Title: Study of Probuphine in Patients With Opioid Dependence
Acronym: PRO-809
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated for reasons not related to efficacy or safety
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-809
Record Dates: First submitted 2008-10-09; First posted 2008-10-15 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependency
Keywords: opioid dependence; opioid addiction; buprenorphine; methadone; heroin; implant; opioid withdrawal; opioid pain medication; suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probuphine (Experimental): buprenorphine implant
  Interventions: Drug: Probuphine (buprenorphine implant)

INTERVENTIONS:
Drug: Probuphine (buprenorphine implant) — Implantable formulation of buprenorphine made of buprenorphine HCl/ethylene vinyl acetate, considered a drug. (4 implants 6-month duration)

SUMMARY:
Buprenorphine (BPN) is an approved treatment for opioid dependence; however, in taking oral tablets, patients experience withdrawal and cravings when the variable BPN levels in the blood are low. Probuphine (buprenorphine implant) is an implant placed just beneath the skin that contains BPN. It is designed to provide 6 months of stable BPN blood levels. This study will test the safety and efficacy of Probuphine in the treatment of patients with opioid dependence. Patients who have completed at least 24 weeks of treatment in the Open-Label, Multi-Center Study of Probuphine in Patients with Opioid Dependence (PRO-807 Study), will be re-treated with Probuphine over an additional 24 weeks.

DETAILED DESCRIPTION:
This is a 6-month, open-label, multi-center extension study. It is estimated that approximately 200 patients will be enrolled at approximately 25 sites in the United States (US). Following completion of either the PRO-807(NCT00630201) or PRO-808 studies, eligible patients will be implanted with Probuphine implants in the opposite arm for the PRO-809 study. Safety, BPN plasma levels, and efficacy measures will be collected during the 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following eligibility criteria:

* Expected to complete 24 weeks of treatment in PRO-807 or PRO-808
* Voluntarily provide written informed consent prior to the conduct of any study-related procedures
* Deemed appropriate for entry into this re-treatment study by the Investigator
* Females of childbearing potential and fertile males must use a reliable means of contraception

Exclusion Criteria:

Patients are not eligible for enrollment if any of the following criteria are met:

* Presence of aspartate aminotransferase (AST) levels ≥ 3 X upper limit of normal and/or alanine aminotransferase (ALT) levels ≥ 3 X upper limit of normal and/or total bilirubin ≥ 1.5 X upper limit of normal and/or creatinine ≥ 1.5 X upper limit of normal, measured at the time of the Week 20 Visit for the previous trial (PRO-807 or PRO-808), or any time less than 5 weeks prior to the Implant Visit.
* Current diagnosis of chronic pain requiring opioids for treatment
* Pregnant or lactating females
* Current use of agents metabolized through cytochrome P450 3A4 (CYP 3A4) such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), and protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* Current history of coagulopathy and anti-coagulant therapy (such as warfarin)
* Current use of benzodiazepines other than physician prescribed use
* Significant medical or psychiatric symptoms, cognitive impairment, or other factors which in the opinion of the Investigator, would preclude compliance with the protocol, patient safety, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in study; and/or any pending legal action that could prohibit participation and/or compliance in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 24 WEEKS

SECONDARY OUTCOMES:
Plasma buprenorphine concentration | 24 WEEKS

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Clinical Research, Inc., North Miami, Florida, United States